CLINICAL TRIAL: NCT06062888
Title: Multi-institutional Phase 2/3 Trial of Fresh Frozen Plasma (FFP) in Patients With Moderate to Severe Traumatic Brain Injury (TBI)
Brief Title: FFP In Traumatic BRAin INjury (FIT-BRAIN) Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Vanderbilt University Medical Center (Other); University of Southern California (Other); Oregon Health and Science University (Other); Medical College of Wisconsin (Other); University of Texas Southwestern Medical Center (Other); University of California, Davis (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hasan Alam, Chair, Department of Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR212312; CDMRP-W81XWH2211106 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Moderate to Severe Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury; Fresh frozen plasma; FFP
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Control vs Experimental Biologic Group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care Control Group
- Standard of Care + FFP (Experimental): Standard of Care + Experimental Treatment
  Interventions: Biological: Fresh Frozen Plasma (FFP)

INTERVENTIONS:
Biological: Fresh Frozen Plasma (FFP) — Standard of Care + 2 units (400-500 ml) of fresh frozen plasma
  Arms: Standard of Care + FFP

SUMMARY:
The goal of this clinical trial is to learn about treatment with fresh frozen plasma (FFP) in individuals with moderate to severe traumatic brain injury. The two main question[s]it aims to answer are:

* Is the FFP treatment safe?
* Does the FFP treatment impact the 24-hour, 3-month and 6-month outcomes, intensive-care free days, mortality, and hospital brain and physical function at discharge. Patients with moderate to severe TBI will randomly receive either:

  * Standard of care treatment
  * Standard of care treatment + 2 units of FFP. Researchers will compare participants receiving standard of care treatment to those receiving experimental fresh frozen plasma (FFP) treatment to see if the FFP is safe and beneficial to participant outcomes.

DETAILED DESCRIPTION:
The two units of fresh frozen plasma will consist of 400-500 ml. The 24-hour, 3-month and 6-month outcome measures include hemorrhagic progression of contusion (HPC) measured on 24-hour follow-up CT scan, the Disability Rating Score (DRS), 24-hour Glasgow Coma Scale (GCS) and the 3-month and 6-month Extended Glasgow Outcome Score (GOS-E).

A third sub aim of the trial is to establish peripheral blood biomarkers, and radiographic features on the initial cross- sectional imaging, that could identify the optimal target population and predict the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 65 years
2. Moderate to severe TBI: GCS 3-12
3. Cerebral trauma confirmed on the initial CT scan with radiographic findings consistent with Brain Injury Guidelines category 3 (BIG 3).
4. The potential participant's wallet, when present, was examined and no power of attorney related to blood product administration was identified.

Exclusion Criteria:

1. Persons with a known history of adverse reaction to plasma products.
2. Persons with a known history of congestive heart failure, renal failure, liver failure, or severe respiratory dysfunction requiring home use of supplemental oxygen.
3. Persons who are currently incarcerated.
4. Persons with inadequate venous access.
5. Treatment cannot start within 1 hour of arrival at the hospital.
6. The time of injury is unknown.
7. Non-survivable injuries in the estimation of the attending trauma and/or neurosurgeon.
8. Interfacility transfers
9. Class 3 hemorrhagic shock
10. Persons with known "do not resuscitate" orders prior to randomization
11. Persons who refuse the administration of blood products
12. Persons with a research "opt out" bracelet
13. Persons who require FFP for any other indication (e.g., reversal of coagulopathy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Extended Glasgow Outcome Scale (GOS-E) | 3 months
  Scoring values range from 1 to 8 with higher scores representing a better outcome. 1 indicates death, 2 indicates a vegetative state, 3 or 4 indicates severe disability, 5 or 6 indicates moderate disability, and 7 or 8 indicates good recovery.

SECONDARY OUTCOMES:
Hemorrhagic progression of the contusion (HPC) | The first 24 hour post-injury
  We will quantify HPC as the change in volume of the largest contiguous brain lesion in mm. This will be measured through a comparison of the initial and the follow-up CT scan.
Disability Rating Scale (DRS) | Discharge or day 7 of the hospital stay and 3 months post-injury
  This scale includes eight categories: A. Eye opening (0-5), B. Communication ability (0-4), C. Motor response (0-5), D. Feeding - cognitive ability only (0-3), E. Toileting - cognitive ability only (0-3), F. Grooming - cognitive ability only (0-3), G. Level of functioning - physical, mental, emotional or social function (0-5) and H. "Employability" - a full time worker, homemaker, or student (0-3). Higher scores in each category mean a worse outcome.

OTHER OUTCOMES:
Disability Rating Scale (DRS) | 6 months post-injury
  This scale includes eight categories: A. Eye opening (0-5), B. Communication ability (0-4), C. Motor response (0-5), D. Feeding - cognitive ability only (0-3), E. Toileting - cognitive ability only (0-3), F. Grooming - cognitive ability only (0-3), G. Level of functioning - physical, mental, emotional or social function (0-5) and H. "Employability" - a full time worker, homemaker, or student (0-3). Higher scores in each category mean a worse outcome.
Extended Glasgow Outcome Scale (GOS-E) | 6 months post-injury
  Scoring values range from 1 to 8, with higher scores representing a better outcome. 1 indicates death, 2 indicates a vegetative state, 3 or 4 indicates severe disability, 5 or 6 indicates moderate disability, and 7 or 8 indicates good recovery.
Time to treatment | The first 24 hours post-injury
  Time to treatment measured in hours and minutes.
Contusion volume | The first 24 hours post-injury
  Total contusion volume measured in mm3
Non-contiguous contusions | The first 24 hours post-injury
  Count of non-contiguous contusions
Glasgow Coma Scale (GCS) | The first 24 hours post-injury
  This scale uses three behavior categories to measure response with larger numbers and total score representing a better outcome. They are: Eye opening response (4-1), Best verbal response (5-1) and Best motor response (6-1). Of the total score 15=Best response, 8 or less = Comatose client and 3=Totally unresponsive.
TBI severity sub-stratification using the Glasgow Coma Scale (GCS) | The first 24 hours post-injury
  his scale uses three behavior categories to measure response with larger numbers and total score representing a better outcome. They are: Eye opening response (4-1), Best verbal response (5-1) and Best motor response (6-1). Of the total score 15=Best response, 8 or less = Comatose client and 3=Totally unresponsive. (GCS 9-12) = moderate and (GCS 3-8)=severe

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Liggett MR, Lashley S, Gill NP, Scholtens DM, Dawood ZS, Alam HB. Plasma therapy for traumatic brain injury: Rationale for a prospective randomized trial. Transfusion. 2024 Jul;64(7):1362-1371. doi: 10.1111/trf.17928. Epub 2024 Jun 28. No abstract available. PMID 38940059
- [Background] Joseph B, Obaid O, Dultz L, Black G, Campbell M, Berndtson AE, Costantini T, Kerwin A, Skarupa D, Burruss S, Delgado L, Gomez M, Mederos DR, Winfield R, Cullinane D; AAST BIG Multi-institutional Study Group. Validating the Brain Injury Guidelines: Results of an American Association for the Surgery of Trauma prospective multi-institutional trial. J Trauma Acute Care Surg. 2022 Aug 1;93(2):157-165. doi: 10.1097/TA.0000000000003554. Epub 2022 Mar 28. PMID 35343931
- [Derived] Jin G, Liggett MR, Ho JW, Dawood ZS, Chtraklin K, Diaz D, Alam HB. Plasma treatment is associated with decreased brain lesion and resuscitation requirements after traumatic brain injury in a swine model of prolonged damage-control resuscitation. J Trauma Acute Care Surg. 2024 Dec 1;97(6):954-960. doi: 10.1097/TA.0000000000004457. Epub 2024 Oct 15. PMID 39733294